CLINICAL TRIAL: NCT00875966
Title: Comparative, Randomized, Single-Dose, 2-Way Crossover Bioavailability Study of Eon and Pfizer Inc. (ZITHROMAX) 200mg/5mL Azithromycin Suspension Following a 600mg Dose in Healthy Adult Volunteers Under Fed Conditions
Brief Title: Comparative Bioavailability Study of Azithromycin 200mg/5mL Suspension Following a 600mg Dose Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D., VP Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA17045
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-04

CONDITIONS: Infections
MeSH Terms: conditions — Infections | interventions — Azithromycin; Suspensions

ARMS (2):
- 1 (Experimental): Azithromycin for oral suspension 200mg/5mL
  Interventions: Drug: Azithromycin for Oral Suspension 200mg/5mL Eon Pharma, LLC
- 2 (Active Comparator): Zithromax (azithromycin for oral suspension) 200mg/5mL
  Interventions: Drug: Zithromax (azithromycin for oral suspension) 200mg/5mL Pfizer

INTERVENTIONS:
Drug: Azithromycin for Oral Suspension 200mg/5mL Eon Pharma, LLC
  Arms: 1
Drug: Zithromax (azithromycin for oral suspension) 200mg/5mL Pfizer — Subjects randomized to Zithromax received a single oral dose of Zithromax 600mg (15mL), administered with 240mL of water under fed conditions
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence of Azithromycin 200mg/5mL oral suspension.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant findings on physical exam, medial history or laboratory tests on screening

Exclusion Criteria:

* Positive test for HIV or hepatitis B and C
* Treatment for Drug or alcohol abuse
* Any other important criteria in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-08; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 37 days